CLINICAL TRIAL: NCT04347330
Title: Cardiovascular Risk Reduction in Atrial Fibrillation Trial
Acronym: CRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Heart Health Research Center (Other); The George Institute for Global Health, China (Other); The George Institute for Global Health, Australia (Other); Fukuoka University (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-005
Record Dates: First submitted 2020-03-29; First posted 2020-04-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: Intensive blood pressure control; Cardiovascular events
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive BP Control (Experimental): Participants randomized into the Intensive BP Control arm will have a goal of home SBP <120mmHg. For most participants in the Intensive Group, a two- or three-drug regimen should be initiated at randomization. Following the randomization visit, addition of another drug or medication dose titration is indicated if home SBP is ≥120 mmHg. Monthly visits will continue in the Intensive Group until home SBP <120 mmHg or no more titration planned. If the home SBP is not <120 mmHg at the every 6-month visit, then an antihypertensive drug from a class different from what is being taken should be added, rather than up-titration the dosage of previous drugs, unless there are compelling reasons against this practice.
  Interventions: Drug: Intensive BP Control
- Standard BP Control (Active Comparator): Participants randomized into the Standard BP Control arm will have a goal of home SBP <135mmHg. The Standard BP protocol is designed to achieve a home SBP of 130-134 mmHg in as many participants as possible. Following the randomization visit, medication dose titration or addition of another drug is indicated if home SBP ≥135 mmHg. Monthly visits will continue in the Standard Group when home SBP ≥155 mmHg. Down titration (a reduction of the dose or number of antihypertensive drugs) should be carried out if the home SBP is <125 mmHg.
  Interventions: Drug: Standard BP Control

INTERVENTIONS:
Drug: Intensive BP Control — Participants in the Intensive group have a goal of home SBP <120 mm Hg. The CRAFT BP treatment protocol is flexible in terms of the choice and doses of antihypertensive medications, but there should be preferences among the drug classes, based on CVD outcome trials results and current guidelines. Use of once-daily antihypertensive agents will be encouraged unless alternative frequency is indicated/necessary. Combination of different classes of agents are encouraged to achieve the home SBP goal. Medications will not be provided by the CRAFT study.
  Other Names: Control of home SBP to a target of 120mmHg
  Arms: Intensive BP Control
Drug: Standard BP Control — Participants in the Standard group has a goal of home SBP <135 mmHg. The same principle of BP treatment in the Intensive BP arm will be used for the Standard BP arm. Medications will not be provided by the CRAFT study.
  Other Names: Control of home SBP to a target of 135mmHg
  Arms: Standard BP Control

SUMMARY:
Atrial fibrillation (AF) is a serious public health problem because of its increasing incidence and prevalence in the aging population. AF is associated with elevated risks of death, stroke, coronary event, heart failure, cognitive decline, and chronic kidney disease. To identify preventive interventions for major cardiovascular events beyond effective anticoagulation should be a major priority in the treatment of AF patients. The CRAFT study is a 2-arm, multicenter, randomized clinical trial designed to test whether intensive blood pressure control will reduce the risk of major cardiovascular events in AF patients.

DETAILED DESCRIPTION:
The CRAFT trial will include approximately 1675 AF patients with home SBP 125-154 mmHg and at least another cardiovascular risk factor. The trial aims to compare the effects of randomization to a treatment program of an intensive SBP goal (target home SBP <120mmHg) with randomization to a treatment program of a standard goal (target home SBP <135mmHg). The primary hypothesis is that cardiovascular event rates will be lower in the intensive arm. Participants will be recruited over a 4-year period at approximately 100 to 150 clinical centres and the first patient will be followed for up to 5 years.

ELIGIBILITY:
Screening and Run-in Assessment

All patients with documented AF (paroxysmal, persistent) and standard office SBP 140-179 mmHg if not on BP-lowering drugs or 125-164 mmHg with BP-lowering drugs, will be screened for inclusion into the run-in assessment phase.

The run-in assessment is for 2 weeks. In the run-in phase, patients should be treated according to guideline recommendation, with combined antihypertension agents. Patients should also be guided to measure and upload HBPM measurements correctly. BP measurements (3 readings in the morning and 3 readings in the evening) are required to be uploaded every day for a week before the end of run-in assessment. Patients with average home SBP 125-154 mmHg during the run-in assessment are considered eligible for study inclusion. If home SBP ≥155 mmHg or <125 mmHg at the time of run-in assessment, another 2 weeks run-in phase can be extended, during which time antihypertensive drugs can be titrated according to the BP lowering algorithm used in this study.

Inclusion Criteria

1. Adults, ≥18 years old
2. Documented AF: persistent atrial fibrillation or at least two episodes of intermittent atrial fibrillation in the previous 6 months.
3. Home SBP 125-154 mmHg, defined as average of all SBP readings (at least 3 readings 1 min apart in the morning before taking antihypertensive drugs and evening before going to sleep) during the run-in assessment.
4. One or more cardiovascular risk factors: (1) Prior history of thromboembolism: defined as any of the following criteria: a) ischemic stroke; b) transient ischemic attack (TIA); c) systemic embolism (SE); (2) Diabetes mellitus (DM): defined as any of the following criteria: a) use of oral hypoglycemic drugs or insulin; b) random blood glucose values ≥11.1 mmol/L in the presence of classic symptoms of hyperglycemia; c) fasting plasma glucose values ≥7.0 mmol/L; d) two-hour plasma glucose values ≥11.1 mmol/L during an oral glucose tolerance test; e) HbA1C values ≥6.5%; (3) Coronary artery disease or Peripheral artery disease: defined as any of the following criteria: a) Previous myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), carotid endarterectomy (CE), carotid stenting; b) Peripheral artery disease (PAD) with revascularization; c) Acute coronary syndrome with or without resting ECG change, ECG changes on a graded exercise test, or positive cardiac imaging study; d) At least a 50% diameter stenosis of a coronary, carotid, or lower extremity artery; e) Abdominal aortic aneurysm ≥5 cm with or without repair; (4) Chronic kidney disease (CKD): defined as estimated glomerular filtration rate (eGFR) 30-59ml/min/1.73m2 based on the latest lab value within the past 6 months; (5) Age ≥65 years old

Exclusion Criteria

1. Successful AF ablation (no documented recurrence of AF, atrial flutter, or atrial tachycardia lasting >30s)
2. Moderate-to-severe mitral stenosis, or mechanical heart valve replacement
3. Home SBP ≥145 mmHg while already taking ≥4 full dose BP lowering agents, indicating resistant hypertension or poor adherence.
4. Unable to upload home BP readings for at least 5 days during the run-in assessment.
5. An indication for a specific BP lowering medication (e.g., beta-blocker following acute myocardial infarction) that the person is not taking, without evidence of intolerance. The screenee should be on the appropriate dose of such medication before assessing whether he/she meets the CRAFT inclusion criteria.
6. Known secondary cause of hypertension that causes concern regarding safety of the protocol.
7. One minute standing SBP < 110 mm Hg. Not applicable if unable to stand due to wheelchair use.
8. Diagnosis of polycystic kidney disease
9. Glomerulonephritis treated with or likely to be treated with immunosuppressive therapy
10. eGFR <30 mL/min/1.73m2 or end-stage renal disease (ESRD)
11. Cardiovascular event or procedure (as defined above as Coronary artery disease or Peripheral artery disease for study entry) or hospitalization for unstable angina within last 3 months
12. Heart failure with reduced left ventricular ejection fraction (< 40%), or New York Heart Association Class III-IV
13. Individuals who have been previously diagnosed with dementia by their physicians
14. A medical condition likely to limit survival to less than 3 years, or a cancer diagnosed and treated within the past two years that, in the judgment of clinical study staff, would compromise a participant's ability to comply with the protocol and complete the trial.
15. Any factors judged by the investigator to be likely to limit adherence to interventions. For example, active alcohol or substance abuse, significant memory or behavioural disorder.
16. Currently participating in another clinical trial (intervention study). Note: Patient must wait until the completion of his/her activities or the completion of the other trial before being screened for CRAFT.
17. Living in the same household as an already randomized CRAFT participant
18. Any organ transplant
19. Unintentional weight loss > 10% in last 6 months
20. Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1675 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite cardiovascular outcomes | 5 years
  a hierarchical composite of cardiovascular death, number of strokes, time to first stroke, number of MI, time to first MI, number of HF, and time to first HF

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Time to all deaths.
Main secondary cardiovascular outcomes | 5 years
  Time to the first occurrence of the components of the primary outcome: cardiovascular Death, stroke, myocardial infarction, hospitalization for heart failure.
Main secondary renal outcomes | 5 years
  Time to the first occurrence of chronic kidney disease progression or incident albuminuria.
Change of the health state utility | 5 years
  Change of the health state utility (measured by the EuroQoL Group 5-Dimension Self-Report questionnaire from baseline to the end of the study.
Change of the self-report depression | 5 years
  Change of the depression (measured by the Patient Health Questionnaire-9) from baseline to the end of the study.
Change of the self-report anxiety | 5 years
  Change of the anxiety (measured by the Zung Self-rating Anxiety Scale) from baseline to the end of the study.
Change of the concern of falling | 5 years
  Change of the concern of falling (measured by the Short Fall Self-Efficacy Scale International) from baseline to the end of the study.
Change of the frailty | 5 years
  Change of the frailty (measured by the 5-item FRAIL scale) from baseline to the end of the study.

OTHER OUTCOMES:
Major bleeding | 5 years
  Time to the first major bleeding (ISTH definition).
Peripheral arterial disease | 5 years
  Time to the first peripheral arterial disease, including systemic embolism, carotid and peripheral revascularization, abdominal aortic aneurysm repair, and other objectively defined PAD events.
Coronary revascularization | 5 years
  Time to the first occurrence of percutaneous coronary intervention or coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Doctor, Principal Investigator — Beijing Anzhen Hospital; Craig S Anderson, Doctor, Principal Investigator — The George Institute for Global Health, China; Heart Health Research Centre; Jianzeng Dong, Doctor, Principal Investigator — Beijing Anzhen Hospital; The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang C, Wang Z, Du X, Wang Y, Gao M, Jia Z, Chai Z, Yang Z, Wang C, He L, Hu R, Lv Q, Wu J, Li X, Jia C, Han R, Arima H, Wang X, Neal B, Rodgers A, Hillis GS, Patel A, Li Q, Dong J, Anderson CS, Ma C. Protocol for a randomized controlled trial of intensive blood pressure control on cardiovascular risk reduction in patients with atrial fibrillation: Rationale and design of the CRAFT trial. Am Heart J. 2024 Dec;278:33-40. doi: 10.1016/j.ahj.2024.08.008. Epub 2024 Sep 7. PMID 39182902